CLINICAL TRIAL: NCT07142057
Title: An Observational Study on the Impact of the 23-valent Pneumonia Vaccine on the Incidence of Pulmonary Infection and Survival in Lung Cancer Patients
Brief Title: An Observational Study on the Impact of the 23-valent Pneumonia Vaccine on Lung Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yalei Zhang, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 23V-PNEUMO-LC
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: LUNG CANCER
MeSH Terms: conditions — Lung Neoplasms | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccination group: Lung cancer patients receive 23-valent pneumonia vaccine
  Interventions: Biological: 23-valent pneumococcal vaccine
- Unvaccinated group: Lung cancer patients have not received the 23-valent pneumococcal vaccine

INTERVENTIONS:
Biological: 23-valent pneumococcal vaccine — Receive the 23-valent pneumococcal vaccine; Do not receive the 23-valent pneumococcal vaccine
  Groups: Vaccination group

SUMMARY:
To evaluate the impact of the 23-valent pneumonia vaccine on the incidence of pulmonary infection and survival in lung cancer patients, and to explore its preventive effect and safety in the lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >=18 years of age;
2. Histological diagnosis of NSCLC, including both non-small cell lung cancer and small cell lung cancer, regardless of whether they are in the early, locally advanced stage or advanced stage, and regardless of whether they have received surgery, radiotherapy, chemotherapy or other treatments;
3. Never received pneumococcal vaccine

Exclusion Criteria:

Patients having other factors that preventing researchers from enrollment them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients can receive or not receive the 23-valent pneumococcal vaccine
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of pneumonia at 12 months | 12 months
  During the 12-month follow-up period, the incidence of pulmonary infection in lung cancer patients was evaluated through regular clinical examinations, imaging tests, and laboratory tests.
Incidence of pneumonia | 24 months
  The proportion of lung cancer patients who developed pneumonia during the study period.

SECONDARY OUTCOMES:
Survival rate | 5 years
  The survival rate of lung cancer patients within a specific time period (such as 1 year, 2 years, or 5 years).

OTHER OUTCOMES:
Lung cancer-related complications | 5 years
  The incidence of complications related to lung cancer (such as respiratory failure, infection, etc.).
Length of hospital stay | 5 years
  Record the number of days of hospitalization for patients hospitalized due to lung infection.
Hospitalization rate | 5 years
  The proportion of patients hospitalized due to pneumonia or other related complications.
Antibiotic usage | 5 years
  This includes the types, dosages, and durations of antibiotic usage, etc
Quality of life of lung cancer patients | 5 years
  Specific quality of life assessment scales are used, such as standardized quality of life assessment tools (such as EORTC QLQ-C30) to evaluate the quality of life of patients.
Immune response | 5 years
  The immune response (such as antibody levels) of patients after vaccination is evaluated through serological testing.
Adverse reactions after vaccination | 30 days
  Observe whether patients who receive the 23-valent pneumococcal vaccine experience adverse reactions after vaccination, such as fever, redness, swelling and pain at the injection site, headache, dizziness, etc.